CLINICAL TRIAL: NCT05487833
Title: Comparison of Insulin and Standard Management in Hypertriglyceridemic Acute Pancreatitis in Patients Without Diabetes
Brief Title: Insulin and Standard Management in Hypertriglyceridemic Acute Pancreatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jakob Gubensek, Principal investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: InzulinHTGAP
Record Dates: First submitted 2022-04-06; First posted 2022-08-04 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Hypertriglyceridemia; Acute Pancreatitis
MeSH Terms: conditions — Hypertriglyceridemia; Pancreatitis | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insulin (Experimental)
  Interventions: Biological: insulin
- standard management (Placebo Comparator)
  Interventions: Other: standard treatment

INTERVENTIONS:
Biological: insulin — 5% glucose in 0.9% NaCl with 4 IU of short acting insulin per 500 ml added, infused at a rate determined by the treating physician, treatment duration: 18 hours
  Arms: insulin
Other: standard treatment — infusion of a balanced solution, infused at a rate determined by the treating physician, treatment duration: 18 hours
  Arms: standard management

SUMMARY:
To compare the efficacy of infusion containing insulin and infusion without insulin on reduction of triglycerides in acute hypertriglyceridemic pancreatitis

ELIGIBILITY:
Inclusion Criteria:

* acute pancreatitis
* triglycerides > 15 mmol/l

Exclusion Criteria:

* diabetes on peroral therapy or insulin
* blood glucose > 11 mmol/l
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
%triglyceride reduction | after 18 hours of treatment
  change in triglycerides, expressed as % of initial value

SECONDARY OUTCOMES:
incidence of hypoglycemia | during treatment with insulin, up to day 5

IPD SHARING:
Plan to Share IPD: Yes
deidentified IPD that underlie results in a publication will be available from the corresponding author on reasonable request